CLINICAL TRIAL: NCT04226820
Title: Peripheral Vascular REactivity and Muscular Oxygenation in Diabetes Mellitus
Acronym: PREMOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B670201940995
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Vascular Complications; Mitochondrial Diseases
Keywords: diabetes mellitus; muscular oxygenation; vascular function
MeSH Terms: conditions — Diabetes Mellitus; Mitochondrial Diseases | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: Participants are divided into 3 groups based on their diagnosis: diabetes mellitus type 1, diabetes mellitus type 2, and healthy persons. Each participant (independent of group) will have the same examinations. There is no retesting of the same participant in other conditions.
Masking Description: There is no masking because the participant knows his diagnosis. Besides, the investigator checks the blood sugar at different times during the examinations, so also the investigator is not blinded. In this study, blinding would have no additional value.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participant (Experimental): Participants are divided into 3 groups based on their diagnosis: diabetes mellitus type 1, diabetes mellitus type 2, and healthy persons. Each participant (independent of group) will have the same examinations. There is no retesting of the same participant in other conditions.
  Interventions: Other: examination: blood pressure assessment; Other: examination: Flow Mediated Dilatation (FMD)-test; Other: examination: handgrip exercise test with Near infrared spectroscopy (NIRS)-monitoring; Other: examination: measurement of glucose by a finger prick

INTERVENTIONS:
Other: examination: blood pressure assessment — blood pressure measurement for 30 minutes, dominant side
Other: examination: Flow Mediated Dilatation (FMD)-test — Flow Mediated Dilatation (FMD)-test for measuring the endothelial functionality
Other: examination: handgrip exercise test with Near infrared spectroscopy (NIRS)-monitoring — participant does a maximal exercise test by a handgrip strength test with simultaneously monitoring of the muscular oxygenation
Other: examination: measurement of glucose by a finger prick — follow-up of blood sugar (glucose) during examinations by a finger prick

SUMMARY:
Oxygen is required for an optimal muscle function. In patients with diabetes mellitus, hyperglycemia can cause vascular complications. The endothelium (inter layer of the blood vessels) can be damaged leading to a reduced oxygen flow towards the muscle cells. Besides, it is possible that mitochondrial dysfunction is occuring leading to reduced extraction of oxygen.

Both conditions will lead to a reduced flow of oxygen towards the muscle and this can have impact on the production of energy necessary for optimal functioning.

In this study, the investigators will examine the functionality of the blood vessels (1) and the uptake of oxygen into the muscles (2) in patients with diabetes mellitus type 1 and type 2 (with and without vascular complications) compared to healthy persons.

DETAILED DESCRIPTION:
The investigators plan to recruit in total 125 participants who will be divided into 3 main groups: (I) diabetes mellitus type 1 (with (a) or without (b) vascular complications), (II) diabetes mellitus type 2 (with (a) or without (b) vascular complications), and (III) healthy persons. Diabetes mellitus will be defined by the guidelines of the American Diabetes Association (ADA).

The examinations for this study consist of a blood pressure assessment, Flow Mediated Dilatation (FMD)-measurement, and a handgrip exercise test. The protocol will take approximately 2 hours.

The investigator who performs the FMD-test followed a course and passed thorough evaluation.

The blood pressure assessment will be continuously for 20 minutes to avoid large bias.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age 18-85 years old
* diabetes mellitus type 1 or type 2 (with or without vascular complications, healthy participants

Exclusion Criteria:

* other types of diabetes mellitus than type 1 or type 2
* alcohol abuse
* active cancer
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilatation (FMD)-test | 20 minutes, at study-day (participants have to come only once, no follow-up, no re-testing)
  flow mediated dilatation test
Near-infrared spectroscopy during exercise | 30 minutes, at study-day (participants have to come only once, no follow-up, no re-testing)
  analysis of changes in oxygenated blood during exercise
exercise test wilt hand held dynamometer | 30 minutes, at study-day (participants have to come only once, no follow-up, no re-testing)
  analysis of strength and exercise capacity

SECONDARY OUTCOMES:
Blood pressure analysis | 20 minutes, at study-day (participants have to come only once, no follow-up, no re-testing)
  measurement of basal blood pressure (systolic and diastolic)

CONTACTS AND LOCATIONS:
Overall Officials: Samyah Shadid, Prof. dr., Principal Investigator — University hospital of Ghent and University of Ghent
Locations (1):
- University Gent, Rehabilitation Sciences, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No